CLINICAL TRIAL: NCT02870257
Title: Effects of Overload Progressive in the Treatment of Shoulder Impingement Syndrome Associated With Scapular Dyskinesis: a Randomized Controlled Trial
Brief Title: Effects of Overload Progressive in the Treatment of Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, André Serra Bley, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.487.198
Record Dates: First submitted 2016-08-04; First posted 2016-08-17 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive overload strengthening group (Experimental): Strengthening protocol with progressive load
  Strengthening muscle exercises for the shoulder and scapular with progressive increase of load during 10 weeks (20 sessions)
  Interventions: Other: Strengthening protocol with progressive load
- Strengthening group (Active Comparator): Strengthening protocol without progressive load
  Strengthening muscle exercises for the shoulder and scapular without increase of load (minimal load) during 10 weeks (20 sessions)
  Interventions: Other: Strengthening protocol without progressive load

INTERVENTIONS:
Other: Strengthening protocol with progressive load — Strengthening protocol for scapular and shoulder muscles
  Arms: Progressive overload strengthening group
Other: Strengthening protocol without progressive load — Strengthening protocol for scapular and shoulder muscles
  Arms: Strengthening group

SUMMARY:
Seventy subjects with shoulder impingement syndrome associated with scapular dyskinesis will be recruited and randomized into two groups of treatment. The group "a" will receive a strenghtening protocol with progressive overload during 20 sessions and group "b" will receive the same protocol with minimal load, without change during the 20 sessions. The primary outcomes measures will be pain, function, quality of life, global impression of recovery. The change will be measure from baseline at 10 weeks (after 20 sessions), 3 and 6 months (follow-up). The secundary outcomes will be disability, quality of life measure by other instruments, shoulder muscle strength and scapular 3d kinematic variables. For these data, change will be measure from baseline at 10 weeks (after 20 sessions).

ELIGIBILITY:
Inclusion Criteria:

* People with diagnosis shoulder impingement syndrome or supraspinatus/rotator cuff tendinopathy or subacromial bursitis
* shoulder pain for more than 4 months, at least 4 points of pain in 0-10 NPRS
* at least 130° shoulder active elevation
* 3 or more positive of 5 physical examination tests (painful arc, external rotation resistence, Neer, empty can (Jobe) and Hawkins-Kennedy
* positive dynamic scapular dyskinesis in clinical observation

Exclusion Criteria:

* Referred pain from vertebral spine
* previous shoulder, elbow or neck surgery
* complete rotator cuff tear (positive drop arm sign or substantial shoulder elevation or rotation weakness)
* neoplastic or neurological disorders
* previous fracture or dislocation injury (shoulder, humerus, clavicle)
* adhesive capsulitis signs
* inflammatory diseases
* specific treatment for the shoulder in the previous four months (injection, physiotherapy)
* using drugs in the previous week
* inability to understand portuguese language

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Numeric pain rating scale (0-10) | baseline, 10 weeks, 3 months and 6 months
Change in SPADI (Shoulder Pain and Disability Index) Questionnaire (0-100) | baseline, 10 weeks, 3 months and 6 months
Change in ASES (American Shoulder and Elbow Surgeons) Questionnaire (0-100) | baseline, 10 weeks, 3 months and 6 months

SECONDARY OUTCOMES:
Disabilities | Change from baseline at 10 weeks
  DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire (0-100)
Quality of life | Change from baseline at 10 weeks
  WORC (The Western Ontario Rotator Cuff Index) Questionnaire (0-100)
Muscle Strength | Change from baseline at 10 weeks
  Shoulder internal rotation, external rotation, adduction and abduction muscles measured by handheld dynamometer
Scapular kinematic | Change from baseline at 10 weeks
  3D data of scapula at 30, 60, 90 and 120° of shoulder abduction
Global impression of recovery | Change from baseline at 10 weeks, 3 months and 6 months
  GPE (global perceived effect) scale (-5 to +5)

CONTACTS AND LOCATIONS:
Overall Officials: André S Bley, Msd, Principal Investigator — University of Nove de Julho
Locations (1):
- UNINOVE, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided